CLINICAL TRIAL: NCT04901182
Title: The Effect of Nutrition-dense, Blenderized Enteral Nutrition From Natural Ingredients on Swallowing Capacity to Prevent Suffocation in the Elderly by Using Flexible Endoscopic Examination of Swallowing (FEES)
Brief Title: Nutrition-dense Smoothie Diets Reduced Dysphagia Risk in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 460/2560(EC3)
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Dysphagia
Keywords: aging; smoothie drink; dysphagia; swallowing capacity
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White sesame soy milk smoothie (WS) (Active Comparator): a formula developed from natural ingredients such as soybean and white sesame
  Interventions: Diagnostic Test: the effect of consuming diets on the swallowing capacity by using Flexible Endoscopic Evaluation of Swallowing (FEES)
- Chicken shitake smoothie (CS) (Active Comparator): a formula developed from natural ingredients such as chicken and shitake mushroom
  Interventions: Diagnostic Test: the effect of consuming diets on the swallowing capacity by using Flexible Endoscopic Evaluation of Swallowing (FEES)
- Ensure (Placebo Comparator): a conventional well-known commercial formula
  Interventions: Diagnostic Test: the effect of consuming diets on the swallowing capacity by using Flexible Endoscopic Evaluation of Swallowing (FEES)

INTERVENTIONS:
Diagnostic Test: the effect of consuming diets on the swallowing capacity by using Flexible Endoscopic Evaluation of Swallowing (FEES) — the effect of consuming white sesame soy milk smoothie (WS), Chicken shitake smoothie (CS) vs. Ensure on the swallowing capacity by using Flexible Endoscopic Evaluation of Swallowing (FEES)

SUMMARY:
The investigators aimed to compare the effect of consuming high protein (23-34% energy ratio) and low carbohydrate (25-38% energy ratio) smoothie formulas vs. consuming Ensure (a conventional well-known commercial formula) on the swallowing capacity by using Flexible Endoscopic Evaluation of Swallowing (FEES) in the elderly people with dysphagia risk.

DETAILED DESCRIPTION:
The investigators aimed to determine the effect of 3 high protein (23-34% energy ratio) and low carbohydrate (25-38% energy ratio) smoothie formulas ((1) white sesame soy milk smoothie (WS), (2) black sesame soy milk smoothie (low carbohydrate, BSLC), and (3) Chicken shitake smoothie (CS); 1 kcal/ml) from natural ingredients as compared with Ensure. The double blind randomized placebo controlled cross-over design study involved 63 subjects aged above 65 years old. They were also divided into asymptomatic (n=32) or symptomatic swallowing difficulty (n=31) group based on self-reported swallowing difficulty symptoms. All subjects assessed five drinks (WS, BSLC, CS vs. Ensure) for sensory testing, product acceptance and marketing survey using questionnaires. Swallowing capacity was determined by using Flexible Endoscopic Examination of Swallowing (FEES) only for each of the three drinks (SW, CS vs. Ensure) in a blinded random sequence.

ELIGIBILITY:
Inclusion Criteria:

* swallowing difficulty group (SSD) who with symptomatic swallowing difficulties or with a history of swallowing difficulties, coughing or choking when eating or drinking or a sign of malnutrition
* control group (WSD) who without a history of swallowing difficulties, coughing or choking when eating or drinking or a sign of malnutrition

Exclusion Criteria:

1. People with chronic illnesses and tube feeding
2. People with anterior bone deformity e.g. facial fracture, sino-nasal or anterior skill-based tumor/surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Level of severity of dysphagia as assessed by a healthcare professional using the FEES | Baseline
  Sum of FEES score from three symptoms consists of premature spillage of material, retention/pooling of material and/or secretion, and entrance of material and/or secretion into the larynx or trachea.
  A healthcare professional evaluated in the five-point scoring system of each symptom.
  FEES score = 5 means there were not exhibit disorder, FEES score = 1 means there were abnormalities at severe level

SECONDARY OUTCOMES:
Premature spillage of material as assessed by a healthcare professional using the FEES | Baseline
  levels of severity of food passed down through the pharynx before swallowing using the five-point scoring system FEES score = 5 means there were not exhibit disorder, FEES score = 1 means there were abnormalities at severe level
Retention/pooling of material and/or secretion as assessed by a healthcare professional using the FEES | Baseline
  levels of severity of food or saliva residue in the vallecular and/or pyriform regions of the pharynx after swallowing using the five-point scoring system FEES score = 5 means there were not exhibit disorder, FEES score = 1 means there were abnormalities at severe level
Entrance of material and/or secretion into the larynx or trachea; presence/absence of reflex cough as assessed by a healthcare professional using the FEES | Baseline
  levels of severity of food passes through the larynx or trachea when swallowed with or without the cough reflex using the five-point scoring system FEES score = 5 means there were not exhibit disorder, FEES score = 1 means there were abnormalities at severe level

CONTACTS AND LOCATIONS:
Overall Officials: Korapat Mayurasakorn, MD., Principal Investigator — Doctor in Family Medicine
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mongkolsucharitkul P, Pinsawas B, Watcharachaisoponsiri T, Suta S, Pumeiam S, Ophakas S, Surawit A, Ongard S, Keskool P, Thitisakulchai P, Srichayet P, Mayurasakorn K. Evaluating swallowing capacity in older adults with dysphagia: high protein, low carbohydrate smoothie formulas versus commercial formula. BMC Geriatr. 2025 Jul 2;25(1):456. doi: 10.1186/s12877-025-06126-x. PMID 40604458